CLINICAL TRIAL: NCT05427071
Title: Magnetic Marker Localization for Occult Breast Cancer and Target Axillary Dissection in Node-positive Breast Cancer Post-neoadjuvant Chemotherapy
Acronym: MaCTAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Endomagnetics Ltd. (Industry)
Responsible Party: Principal Investigator, Professor Ava Kwong, Daniel CK Yu Professor in Breast Cancer Research, Chief of Breast Surgery Division, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 20-064
Record Dates: First submitted 2022-05-16; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Breast Neoplasm; Chemotherapy Effect
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients received magnetic seeds guided localization of axillary lymph node and breast tumor and superparamagnetic iron oxide-guided sentinel lymph node biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Magnetic seed guided lumpectomy and targeted axillary dissection
  Interventions: Device: Magnetic seed localization

INTERVENTIONS:
Device: Magnetic seed localization — Magnetic seed guided localization

SUMMARY:
The use of neoadjuvant chemotherapy in breast cancer is expanding in the recent decade. Patients with good response to neoadjuvant chemotherapy could benefit from de-escalation of breast and axilla operation. However, breast tumor and involved axillary lymph node should be marked before the commencement of chemotherapy. This could facilitate subsequent operative planning and intraoperative assessment of disease response. This study aims to evaluate the feasibility of magnetic marker localization for non-palpable breast cancer and targeted axillary dissection in patients with node-positive breast cancer following neoadjuvant therapy

DETAILED DESCRIPTION:
Eligible patients will receive ultrasound guided placement of magnetic seeds (Magseed®) within the cortex of the sampled lymph node and epicenter of the breast tumor by radiologists before commencement of neoadjuvant treatment. Chemotherapeutic regimes will be determined by oncologists in charge. During the period of neoadjuvant treatment, patients will be followed up by oncologists and surgeons with clinical assessment of tumor response according to our usual practice. After completion of neoadjuvant chemotherapy, recruited patients will receive mammography and ultrasonography assessment before surgery. Breast conservative surgery with targeted axillary dissection will be offered when feasible. In patients not suitable for breast conservative surgery, mastectomy and targeted axillary dissection with or without immediate breast reconstruction will be offered.

Patient will receive localization of previously marked axillary lymph node and breast tumor and sentinel lymph node biopsy by magnetic means completely, i.e. by the use if magnetic seeds and superparamagnetic iron oxide injection. Radioisotope with Tc-99 is injected prior to operation as backup plan for sentinel lymph node biopsy. The clipped lymph node and sentinel lymph nodes are sent for frozen section analysis. If any of the lymph nodes is positive for malignancy, axillary dissection will be performed. Similarly, the breast tumor will be resected with guidance of magnetometer and specimen mammogram will confirm the presence of tumor and magnetic seeds.

ELIGIBILITY:
Inclusion Criteria:

* All patients with cT1-3N1 invasive ductal carcinoma planned for neoadjuvant chemotherapy and/or target therapy
* mentally competent to give informed consent
* Agreed to proceed with curative operation after chemotherapy and tentatively keen for breast conservative surgery and targeted axillary dissection after neoadjuvant chemotherapy
* Radiologically 1-3 ipsilateral axillary lymph node metastases confirmed by cytology or biopsy

Exclusion Criteria:

* Presence of distant metastasis, inflammatory breast cancers, multi-centric breast cancers
* History of previous ipsilateral axillary surgery or irradiation
* Hypersensitivity to dextran compounds or iron
* Iron overload disease
* Pregnant or lactating patients
* Patients with pacemaker or other implantable metallic devices in chest wall or prosthesis in shoulder
* Mentally incompetent patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful localization of breast tumor and axillary lymph node | At the time of operation
  Successful surgical retrieval of magnetic seed marked breast tumor and axillary lymph node in intraoperative specimen mammogram (in percentage)

SECONDARY OUTCOMES:
Percentage of patients that can avoid axillary lymph node dissection | up to 4 weeks
  Percentage of patients that can achieve nodal pathological complete response after neoadjuvant chemotherapy
Percentage of successful magnetic seed guided lumpectomy | up to 4 weeks
  Percentage of involved or close margins in lumpectomy specimen which require re-excision
Level of satisfaction from surgeons and radiologists | To be filled in by operating surgeons and radiologists at the time of operation or magnetic seeds placement
  Level of satisfaction from surgeons and radiologists which will be determined by the satisfaction questionnaire
5-year local regional recurrence rate | 5-year post-operatively
  5-year ipsilateral breast tumor recurrence rate and/or axillary recurrence rate

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No